CLINICAL TRIAL: NCT06037668
Title: BVR-100 and BES-100 Validation Trial: A Randomized, Double-Blind, Parallel-Group, Controlled Study of Two At-Home Self-Guided Virtual Reality Interventions for Adults With Social Anxiety Disorder.
Brief Title: A Randomized, Controlled Study of Two At-Home Self-Guided Virtual Reality Interventions for Adults With Social Anxiety Disorder.
Acronym: BVR-100-102
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Collaborators: BehaVR LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BVR-100-102
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Social Anxiety Disorder (SAD)
Keywords: Social Anxiety Disorder, Social Phobia
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BVR-100 (Experimental): Experimental at-home VR intervention for the treatment of SAD
  Interventions: Device: BVR-100
- BES-100 (Active Comparator): Active at-home VR intervention comparator
  Interventions: Device: BES-100

INTERVENTIONS:
Device: BVR-100 — Experimental self-guided VR intervention for the treatment of SAD
  Arms: BVR-100
Device: BES-100 — Active at-home VR intervention comparator
  Arms: BES-100

SUMMARY:
This study is to compare two Virtual Reality (VR)-based interventions, BVR-100 and BES-100, for the treatment of Social Anxiety Disorder (SAD).

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, aged 18 or above.
* Subject has English fluency and literacy.
* Subject meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, (DSM-5) criteria for Social Anxiety Disorder
* Subject has a total Liebowitz Social Anxiety Scale (LSAS) score at Screening of ≥ 70.

Exclusion Criteria:

* Subject has significant visual, auditory or balance impairment
* Subject has history of photosensitive epilepsy or seizure disorder
* Subject has history of motion sickness or medical condition predisposing to nausea or dizziness.
* Subject has injuries, inflammation or infection affecting the eyes, ears or face that would make the use of the hardware uncomfortable.
* Subject has, current or lifetime history of meeting DSM-5 criteria for schizophrenia spectrum or other psychotic disorder, bipolar or related disorder, major neurocognitive disorder, neurodevelopmental disorder of greater than mild severity or of a severity that impacts the subject's ability to consent, follow study directions, or otherwise safely participate in the study; posttraumatic stress disorder, major depressive disorder (MDD) with psychotic features, borderline or antisocial personality disorder
* Subject has met DSM-5-based criteria for Alcohol or Substance Use Disorder (other than nicotine or caffeine) within one (1) year prior to Screening.
* Subject has received ketamine, esketamine, arketamine, or psychedelic therapies (eg, psilocybin, methylenedioxymethamphetamine [MDMA]) for MDD or any psychiatric condition within one (1) year prior to Screening.
* In the opinion of the Investigator: (a) study participation may pose a significant or undue risk to the subject; (b) the subject is unlikely to successfully complete all of the requirements of the study per protocol; or (c) study participation may adversely impact the integrity of the data or the validity of the study results.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hayes, PhD, Study Director — Sumitomo Pharma America, Inc.
Locations (6):
- United States (6):
  - CNS Healthcare, Orlando, Florida
  - Curavit Clinical Research, Boston, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - Midwest Research Group, Saint Charles, Missouri
  - Alivation Health, LLC, Lincoln, Nebraska
  - Cedar Clinical Research, Draper, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BVR-100 | BES-100
Started | 28 | 28
Completed | 24 | 27
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other Study Discontinuation Reason | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | BVR-100 | BES-100 | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 25 | 25 | 50
    >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    Female | 15 | 25 | 40
    Male | 10 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    Hispanic or Latino | 2 | 3 | 5
    Not Hispanic or Latino | 22 | 22 | 44
    Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 4 | 6
    White | 20 | 22 | 42
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    United States | 25 | 27 | 52
Baseline Credibility/Expectancy score [Mean (Standard Deviation); unit: units on a scale] — The Credibility/Expectation Questionnaire (CEQ) asks about the improvements that subjects believe will be achieved as a result of treatment, and how believable, convincing, and logical the treatment seems. It contains 6 items (each item is rated on a 1-9 scale). Total CEQ score is calculated for each subject at each visit by taking the sum of score of all 6 items of the scale ranging from 6 to 54. Higher score corresponds to better credibility and expectancy. Population: ITT Population
  units on a scale
    number analyzed (Participants) | 18 | 14 | 32
    (all) | 35.1 (8.13) | 30.2 (6.58) | 32.9 (7.77)
Baseline Credibility score [Mean (Standard Deviation); unit: units on a scale] — The Credibility scale asks about the improvements that subjects think will be achieved as a result of treatment, and how believable, convincing,and logical the treatment seems.It contains three items rated on a 1-9 scale. Higher scores suggest better experience, lower scores suggest poor experience.Credibility score is calculated by taking the sum of score of the first 3 items of the scale ranging from 3 to 27. Population: ITT Population
  units on a scale
    number analyzed (Participants) | 18 | 14 | 32
    (all) | 18 (4.31) | 15.4 (4.57) | 16.9 (4.54)
Baseline Expectancy score [Mean (Standard Deviation); unit: units on a scale] — The Expectancy Score asks about the improvements that subjects feel will be achieved as a result of treatment.It contains three items rated on a 1-9 scale.Higher scores suggest better experience, lower scores suggest poor experience. Expectancy Score is calculated by taking the sum of score of the last 3 items of the scale ranging from 3 to 27. Population: ITT Population
  units on a scale
    number analyzed (Participants) | 18 | 14 | 32
    (all) | 17.1 (4.43) | 14.8 (3.24) | 16.1 (4.06)

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Intervention Credibility Assessed With the Credibility Score, at Baseline
Description: The Credibility/Expectation Questionnaire (CEQ) asks about the improvements that subjects believe will be achieved as a result of treatment, and how believable, convincing,and logical the treatment seems.It contains six items rated on a 1-9 scale. The first three items load onto the credibility factor. Higher scores suggest better experience, lower scores suggest poor experience.Credibility score is calculated by taking the sum of score of the first 3 items of the CEQ scale ranging from 3 to 27.
Time Frame: Baseline
Population: ITT Population who had measurement of Credibility / Expectancy Score completed at Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BVR-100 | BES-100
Number analyzed (Participants) | 18 | 14
units on a scale | 18 (4.31) | 15.4 (4.57)
Statistical Analysis 1: Comparison: BVR-100 vs BES-100; Test type: Superiority; p = 0.1134, Independent t-test — p-values are calculated by independent t-test

2. Primary Outcome: Measurement of Intervention Credibility Assessed With the Credibility Score, at Week 6
Description: as for outcome 1
Time Frame: 6 weeks
Population: ITT Population who had measurement of Credibility / Expectancy Score completed at Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BVR-100 | BES-100
Number analyzed (Participants) | 17 | 17
units on a scale | 18.9 (5.37) | 12.3 (6.56)
Statistical Analysis 1: Comparison: BVR-100 vs BES-100; Test type: Superiority; p = 0.003100, Independent t-test — p-values are calculated by independent t-test

3. Primary Outcome: Measurement of Intervention Credibility Assessed With the Credibility Score, at Week 8
Description: as for outcome 1
Time Frame: 8 weeks
Population: ITT Population who had measurement of Credibility / Expectancy Score completed at Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BVR-100 | BES-100
Number analyzed (Participants) | 15 | 19
units on a scale | 18.7 (6.31) | 13.7 (7.68)
Statistical Analysis 1: Comparison: BVR-100 vs BES-100; Test type: Superiority; p = 0.050300, Independent t-test — p-values are calculated by independent t-test

4. Primary Outcome: Measurement of Intervention Credibility Assessed With Expectancy Score, at Baseline
Description: The Credibility/Expectation Questionnaire (CEQ) asks about the improvements that subjects believe will be achieved as a result of treatment, and how believable, convincing,and logical the treatment seems.It contains six items rated on a 1-9 scale. The final three items load onto the expectancy factor. Higher scores suggest better experience, lower scores suggest poor experience.Expectancy score is calculated by taking the sum of score of the last 3 items of the CEQ scale ranging from 3 to 27.
Time Frame: Baseline
Population: ITT Population who had measurement of Credibility / Expectancy Score completed at Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BVR-100 | BES-100
Number analyzed (Participants) | 18 | 14
units on a scale | 17.1 (4.43) | 14.8 (3.24)
Statistical Analysis 1: Comparison: BVR-100 vs BES-100; Test type: Superiority; p = 0.1178, Independent t-test — p-values are calculated by independent t-test

5. Primary Outcome: Measurement of Intervention Credibility Assessed With the Expectancy Score, at Week 6
Description: as for outcome 4
Time Frame: 6 weeks
Population: ITT Population who had measurement of Credibility / Expectancy Score completed at Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BVR-100 | BES-100
Number analyzed (Participants) | 17 | 17
units on a scale | 15.4 (5.75) | 11.6 (7.14)
Statistical Analysis 1: Comparison: BVR-100 vs BES-100; Test type: Superiority; p = 0.1003, Independent t-test — p-values are calculated by independent t-test

6. Primary Outcome: Measurement of Intervention Credibility Assessed With the ExpectancyScore, at Week 8
Description: as for outcome 4
Time Frame: 8 weeks
Population: ITT Population who had measurement of Credibility / Expectancy Score completed at Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BVR-100 | BES-100
Number analyzed (Participants) | 15 | 19
units on a scale | 15.3 (6.21) | 13.6 (7.47)
Statistical Analysis 1: Comparison: BVR-100 vs BES-100; Test type: Superiority; p = 0.4832, Independent t-test — p-values are calculated by independent t-test

7. Secondary Outcome: Subject Retention Rate at Week 6
Description: Subject retention in each group were assessed by percentage of subjects who remain on the study at Week 6
Time Frame: 6 weeks
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | BVR-100 | BES-100
Number analyzed (Participants) | 24 | 27
percentage of participants | 96 | 100

8. Secondary Outcome: Subject Retention Rate at Week 8
Description: Subject retention in each group were assessed by percentage of subjects who remain on the study at Week 8
Time Frame: 8 weeks
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | BVR-100 | BES-100
Number analyzed (Participants) | 24 | 27
percentage of participants | 96 | 100

9. Secondary Outcome: Summary of Time-on-Task
Description: Time-on-task, averaged over all VR sessions from baseline to Week 8/EOS. Time on task will be automatically recorded by the VR system after each session.
Time Frame: 8 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | BVR-100 | BES-100
Number analyzed (Participants) | 25 | 27
minutes | 4.97 (1.886) | 6.59 (0.359)

ADVERSE EVENTS:
Time Frame: Up to 8 Weeks
Arm/Group | BVR-100 | BES-100
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 3/25 | 0/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BVR-100 (N=25) | BES-100 (N=27)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT06037668/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT06037668/SAP_001.pdf